CLINICAL TRIAL: NCT03067337
Title: Clinical Evaluation Between Zirconia Crowns and Stainless Steel Crowns in Primary Molars Teeth
Brief Title: Evaluation Between Zirconia and Stainless Steel Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Bashaer S. Abdulhadi, PhD Student, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zirconia and SSC
Record Dates: First submitted 2017-01-22; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Tooth Diseases
Keywords: Stainless Steel Crowns; Zirconia Crowns; Aesthetic restorations
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Stainless Steel Crowns (Group A) (Experimental): Groups that received Stainless Steel Crowns
  Interventions: Device: Stainless Steel Crown (Group A)
- Zirconia crowns (Group B) (Experimental): Groups that received Zirconia crowns
  Interventions: Device: NuSmile Zirconia Crowns (Group B)

INTERVENTIONS:
Device: Stainless Steel Crown (Group A) — Full coverage restoration for multi-surface carious teeth
  Other Names: Stainless Steel Crown
  Arms: Stainless Steel Crowns (Group A)
Device: NuSmile Zirconia Crowns (Group B) — Full coverage restoration for multi-surface carious teeth
  Other Names: Zirconia crowns
  Arms: Zirconia crowns (Group B)

SUMMARY:
Introduction and Research Problem:

The aim of this project is to evaluate and compare two full coronal restorations on primary posterior molars over a period of 3, 6 and 12 months in terms of restoration failure, marginal integrity, proximal contact, secondary caries, occlusion and gingival response. The restorations types are Stainless Steel Crowns (SSC) and NuSmile Zirconia Crowns (Nu/ZR).

Materials and Methods:

Children attending the King Abdulaziz University, Faculty of Dentistry (KAUFD) clinics who need restorations will be screened for inclusion criteria till 120 teeth are recruited (60 teeth for SSC restorations and 60 for Nu/ZR restorations). Split mouth technique will be used to ensure equalizing variables for both groups, each patient will have side restored with SSC and the opposite side will be restored with Nu/ZR crowns.

Randomization will be done using Statistical Package for the Social Sciences (SPSS) software version 20.0 (Armonk, New York; International Business Machines Corporation (IBM Corp) for each age group separately with a uniform random variable generation. A simple descriptive statistics will be used for analysis and a T-Tests with Wilcoxon Signed-Rank will be used. Level of significance will be set at (α = 0.05) and level of confidence at (95%).

ELIGIBILITY:
Inclusion Criteria:

* Age group of 4-8 years
* Free of any systemic disease
* Cooperative patient
* At least two matched bilateral carious primary molars
* Minimal of two surfaces of caries in the targeted tooth
* Written consent obtained from the parent/guardian

Exclusion Criteria:

* Any subject that does not fall under the inclusion criteria were excluded.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-08-30 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Gingival health | 3-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe, 1967].
Plaque index | 3-month follow-up
  This parameter was evaluated using a blunt periodontal probe (Double ended probe Williams 1-2-3-5-7-8-9-10 Goldman Fox Flat) according to the Löe and Silness gingival index [Löe,1967].
Restoration failure | 3-month follow-up
  This was clinically evaluated with visual assessment of the restoration, according to the US Public Health Service "USPHS", Alpha criteria rating system [Ryge, 1980].

IPD SHARING:
Plan to Share IPD: No